CLINICAL TRIAL: NCT02596139
Title: Reliability and Validity of the Taiwan-version of Multidimensional Fatigue Inventory and Fatigue Severity Scale
Status: Completed | Type: Observational
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Other Study IDs: 104-0704B
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Fatigue; Taiwan-version Questionnaire
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy people
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions

SUMMARY:
The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.

Fatigue Severity Scale (FSS) contains nine statements that rate the severity of fatigue symptoms. The purposes of this study are to translate fatigue questionnaires of -MFI- and -FSS- to Taiwan-version, and to examine the reliability and validity of the scales.

A hundred adult people without diagnosed physical nor mental disabilities will be recruited. Subjects will fill out the Taiwan-version of MFI, FSS, SF-36 and Pittsburg Sleep Quality Index (PSQI) to establish the validity. Subjects will re-fill the MFI and FSS one week later to evaluate the test-retest reliability.

Another twenty people who are familiar with both English and Chinese will be recruited to evaluate the translation reliability. Subjects will fill out the English version of MFI and FSS and, then, fill out the Taiwan-version of the MFI and FSS with at least ten minutes apart. The translation reliability will be evaluated by paired t test and the intraclass correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* No cognition or mental disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assessing the reliability and validity of Taiwan-version Multidimensional Fatigue Inventory questionnaire | 1 week
Assessing the reliability and validity of Taiwan-version Fatigue Severity Scale questionnaire | 1 week

SECONDARY OUTCOMES:
SF-36 questionnaire | Baseline
  To establish the criterion validity
Pittsburg Sleep Quality Index questionnaire | Baseline
  To establish the criterion validity

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan